CLINICAL TRIAL: NCT07118449
Title: A 26-Week (With 26 Week Extension) Randomized, Multi-Center, Double-Blind Phase 2 Study to Evaluate the Efficacy and Safety of XC001 Gene Therapy as an Adjunct to Coronary Artery Bypass Graft Surgery for Patients With Symptomatic Coronary Artery Disease With Left Ventricular Dysfunction at Risk for Incomplete Revascularization
Brief Title: Epicardial Delivery of XC001 Gene Therapy to Promote Angiogenesis in CAD Patients Undergoing Treatment With CABG
Acronym: EXACT-CABG
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XyloCor Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XC001-1003; 2025-521325-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-17; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Administration of study drug (XC001) at the end of the CABG procedure.
  Interventions: Drug: XC001
- Placebo group (Placebo Comparator): Administration of A195/placebo at the end of the CABG procedure.
  Interventions: Drug: A195/placebo

INTERVENTIONS:
Drug: XC001 — 22 injections will be administered at the end of the CABG procedure as a one time treatment.
  Arms: Treatment group
Drug: A195/placebo — 22 injections of A195/placebo will be administered at the end of the CABG procedure.
  Arms: Placebo group

SUMMARY:
This is a 26-week (with a 26-week extension) multicenter, randomized, double-blind, placebo-controlled Phase 2 study of XC001 versus placebo. Approximately 116 participants who have CAD and have been referred for revascularization by CABG and who have, according to assessment by stress imaging multiple myocardial segments that are substantially ischemic, and that are unlikely to be fully revascularized during CABG for technical reasons, including diffuse atherosclerosis, lack of conduits, or insufficient target vessels.

Patients will be randomized in a 1:1 to XC001 or placebo injections during the final stages of the CABG procedure. Patients will have a baseline CMR at day 4-6 post CABG and additional assessments in the primary study period will be performed on Day 14, and Weeks 4, 12, and 26, (and during the extension period at 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females, age 18 to 80 years, inclusive, at the time of signing the ICF.

  2. Has multivessel epicardial CAD and is clinically indicated for coronary revascularization that is best treated via elective (stand-alone, i.e., not associated with valve surgery) and on-pump CABG at high risk for incomplete revascularization as assessed by local cardiothoracic surgeon and independent Eligibility Review Committee (ERC).

  3. LVEF by standard quantitative imaging technique of 25% to 50%. 4. Anatomical findings on coronary angiography and/or stress imaging that increase the likelihood of incomplete revascularization post-CABG and that supply LV segments determined to be ischemic on pre-operative stress imaging (detailed in the ERC Charter). These include, but are not exclusively:

  a. Diffuse distal coronary artery atherosclerotic disease and/or small coronary target vessels deemed unsuitable for grafting within a major coronary artery b. Multiple segmental lesions along a defined major coronary artery c. In a major coronary artery - "missing vessel" where the vessel is not seen on an angiogram d. Major coronary arteries that are ungraftable due to a long segment of failed stents e. High likelihood of available conduits being insufficient for target lesions in major coronary arteries f. Ischemic regions identified on stress imaging that are not likely to be benefited by CABG (ischemic region greater in size than that portion of myocardium supplied by the target vessel(s) that will likely be successfully grafted). Further detailed in the ERC Charter.

  5. All participants capable of procreation with their partners must agree to use a highly effective and medically accepted method of contraception for 6 months following the study procedure (Day 1) to avoid pregnancy. This is not required of female participants who are either:
  1. Postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to screening. In addition, at least 2 high follicle stimulating hormone (FSH) measurements in the postmenopausal range must be used to confirm a postmenopausal state in women with less than 12 months of amenorrhea and not using hormonal replacement surgery; OR
  2. Surgically sterile (i.e., hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) at least 1 month prior to Screening 6. Female participants agree to not donate oocytes and male participants must agree not to donate sperm for 6 months following administration of investigational protocol.

     7. Capable of providing informed consent and undergoing all the required tests and procedures in the protocol.

     Exclusion Criteria:
* 1. Any of the following:

  1. ST elevation myocardial infarction (STEMI) or cerebral vascular accident within the past 60 days prior to the Screening visit;
  2. Sustained, current systolic blood pressure (BP) less than 90 mmHg or uncontrolled hypertension (systolic BP > 180 mmHg, diastolic BP > 100 mmHg) despite maximal medical treatment;
  3. Current untreated malignant ventricular arrhythmia;
  4. Congestive heart failure (HF) within the last 60 days defined as New York Heart Association Functional Class IV;
  5. Current mitral or aortic valvular heart disease requiring mechanical intervention anticipated during the study period (including percutaneous intervention).

     2. Participants with uncontrolled coagulation disorder (that cannot be corrected by pharmacotherapy).

     3. Participants with documented, active proliferative retinopathy from any cause (ETDRS [Early Treatment Diabetic Retinopathy Study] score >35).

     4. Indication for combination of CABG with any valvuloplasty or valvular replacement and/or arrhythmia surgery (for instance a Cox-maze IV surgical procedure for atrial fibrillation).

     5. Body mass index (BMI) > 45 kg/m2. 6. Hemoglobin < 10 g/dL, absolute neutrophil count < 1.2 × 103 per µL, platelet count < 75,000 per µL, alanine aminotransferase and aspartate aminotransferase > 3 × upper limit of normal (ULN), total bilirubin > 2 × ULN unless the participant has a previously known history of Gilbert's syndrome 7. Diabetic individuals with glycosylated hemoglobin (HbA1c) > 9.5% or with active proliferative diabetic retinopathy.

     8. A history or evidence of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV), active hepatitis B virus (HBV).

     9. Severely immune compromised participants, including participants currently treated with chronic high dose of corticosteroid therapy and/or cytostatic (oncolytic) therapy.

     10. Diagnosis of, or treatment for, any cancer within the last 5 years, except for basal or squamous cell carcinoma or carcinomas in situ where surgical excision was considered curative. Past medical history of cancer is not exclusionary as long as the participant has been disease free for at least 5 years since the time of diagnosis and treatment.

     11. Known hypersensitivity or any other contraindication to the formulation buffer used to suspend the viral vector or contrast agents used in any of the radiographic procedures, or contraindication to general anesthesia.

     12. Pregnancy or currently lactating. 13. Absolute contraindication to CMR: metallic implant (including pacemaker, or implantable cardioverter defibrillator), uncontrolled claustrophobia, severe renal dysfunction (eGFR<30 mL/minute/1.73 m2), or on renal dialysis.

     14. Recurrent or persistent atrial fibrillation with rapid ventricular response (>100 bpm) that precludes the analysis of CMR stress imaging (to assess ischemic burden, cardiac dimensions and cardiac function).

     15. Receiving an investigational intervention or participating in another clinical study within 30 days or within 5 half-lives (whichever is longer) of the drug prior to Screening. An exception may be made if the individual is enrolled in a nontherapeutic observational study (registry) or the observational portion of a therapeutic study where the sponsoring authority authorizes enrollment.

     16. Prior participation in any gene therapy; however, if the study was unblinded or documentation otherwise exists that the participant was randomized to the placebo control group and did not receive active gene transfer agent, the participant may be considered for this study.

     17. Has a serious or unstable medical (including unstable chronic obstructive pulmonary disease under adequate treatment) or psychological condition (including drugs or alcohol abuse) that, in the opinion of the Investigator (with input from the ERC as appropriate), would compromise the participant's safety or successful participation in the study or interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-08-27 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (Day 4-6 CMR) in treated segment(s) comparing XC001 and placebo in CMR imaging parameters at Weeks 12 and 26 post-surgery. | Week 26
  Endpoint at the participant level is the proportion of qualifying segments that improve at 12 and/or 26 weeks as determined by myocardial ischemic burden, as measured by the following:
  * Global and segmental perfusion measured as sum of 32 subsegmental American Heart Association (AHA) LV segments with myocardial ischemia at 12- and 26-weeks follow-up compared to baseline (defined as a subsegment with myocardial ischemia without subendocardial late gadolinium enhancement)
  * Segmental myocardial blood flow measuring extent of ischemic defect in each of 16 (combined subendocardial and subepicardial) AHA LV segments defined as below at 12 and 26 weeks follow-up compared with Baseline:
    * Segment is abnormal if one (subendocardial) or both subsegments are ischemic at Baseline
    * Segment is defined as improved at follow-up if one or both subsegments normalize To qualify for analysis of the primary endpoint, at least 3 of 32 subsegments will have will have to be ischemic on the baseline CMR.

CONTACTS AND LOCATIONS:
Locations (1):
- Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No